CLINICAL TRIAL: NCT02362282
Title: Combined Cognitive and Gait Training
Acronym: CogGait
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to hire qualified personnel to run the study
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7675-R
Record Dates: First submitted 2015-01-29; First posted 2015-02-12 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-09

CONDITIONS: Stroke
Keywords: stroke; walking; cognition; rehabilitation
MeSH Terms: conditions — Stroke | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gait plus cognitive training (Active Comparator): Rehabilitation of walking/gait, combined with rehabilitation of cognitive function
  Interventions: Behavioral: Gait training; Behavioral: cognitive training
- Gait plus arm training (Active Comparator): Rehabilitation of walking/gait, combined with rehabilitation of arm function
  Interventions: Behavioral: Gait training; Behavioral: Arm training

INTERVENTIONS:
Behavioral: Gait training — Treatment will include coordination exercises and over ground gait training for impaired muscle groups and related gait deficits. The therapy will be provided by a clinical physical therapist specializing in rehabilitation for stroke patients, according to established, conventional guidelines. The protocol was used in the investigators' prior studies, and is designed to restore voluntary control of ankle dorsiflexion during swing phase; hip flexion during swing phase, knee flexion at toe-off, knee flexion during swing phase; knee extension before heel strike; knee control during stance phase; pelvic control during stance phase; and whole body balance control during weight shifting. Newly-learned coordinated movements will be integrated into practice of coordinated gait components. Cognitive rehabilitation will begin with the least difficult aspects of attention control, and progress to the more difficult. Home practice and generalization exercises will be assigned.
Behavioral: cognitive training — Cognitive training is designed to enhance attention, intention, executive function, decision making and reaction time. Commercially available computer software will be used, as well as custom cognitive training.
  Arms: Gait plus cognitive training
Behavioral: Arm training — Treatment will include coordination exercises for reaching and grasping. Activities will include movement of shoulder, elbow, wrist and fingers.
  Arms: Gait plus arm training

SUMMARY:
Recent research in gait training for stroke survivors showed that coordinated gait components can be best restored using the following interventions together: coordination exercises, over ground gait training, and body weight supported treadmill training (BWSTT). These results are important because, to the investigators' knowledge, there have been no other reports of the restoration of coordinated gait components for those with persistent gait deficits (> 6 months after stroke). However, a remaining problem was that the restored coordinated gait movements measured in the laboratory did not generalize for many subjects to the everyday environment. The confluence of several factors can cause lack of generalization. First, dual task performance (gait and cognitive attention task) can degrade both gait and attention ability, even in healthy adults. Second, stroke can impair attention. Third, during walking in the everyday environment, attention is required in order to safely process normally occurring stimuli. Therefore, given the success of the new gait training protocol in the lab setting, it is important to address the problems remaining for generalization of the recovered coordinated gait pattern to the everyday environment. The primary hypothesis of this study is that greater gains in gait speed will be produced by combined motor and cognitive training versus motor training alone.

DETAILED DESCRIPTION:
Aim 1, Hypothesis Ia: Comparison of combined motor and cognitive training vs motor training alone. For Aim 1, Hypothesis Ia, this will be a randomized, controlled study. For the two groups, 38 subjects will be enrolled and randomized to either: A) Motor + Cognitive Training; or B) Motor Training alone. Subjects will first be stratified according to coordination and gait deficit severity, as described below. After stratification, the subject will be randomized to one of the two intervention groups for Hypothesis Ia. All the subjects will receive treatment 5 times/week, 3hrs/session, for 12 weeks or for a total of 60 treatment sessions. Group A will receive combined motor and cognitive training; Table 2 (below) shows the graduated approach to providing combined gait and cognitive training. Data collection will be at weeks 1, 6, 12, and 24 (i.e., before, mid-treatment and after treatment, and then 3 months after the end of the treatment protocol. Comparison will be made between the two groups to determine whether there was any additive effectiveness of the cognitive training.

Aim 2, Hypotheses IIa-d: Pre/post-treatment comparisons within Group A, receiving combined motor and cognitive training. For Aim 2, Hypotheses IIa-d, this will be a single cohort pre/post-treatment comparison within Group A receiving combined motor and cognitive training.

Aim 3, Hypotheses IIIa-d: Pre/post-treatment comparisons within Group B, receiving motor training alone. For Aim 3, Hypotheses IIIa-d, this will be a single cohort pre/post-treatment comparison within Group B, receiving motor training alone.

ELIGIBILITY:
Inclusion Criteria:

Stroke Survivor inclusion/exclusion criteria Inclusion Criteria

* Cognition sufficiently intact to give valid informed consent to participate. *
* Sufficient endurance to participate in rehabilitation sessions.
* Ability to follow 2 stage commands.
* Medically Stable
* Age > 21 years.
* Impaired ambulation as follows: inability to flex the knee and ankle in the sagittal plane, in a normal manner so the foot clears the floor; inability to control normal knee angle during single limb weight bearing during stance phase.
* At least 6 months post stroke.

Able-bodied Inclusion criteria

* Criteria to be included is that they should be healthy with no history of a neurological disease or orthopedic impairment.**
* Not Pregnant.
* No Claustrophobia (only for the sub-sample asked to undergo fMRI.)
* No counterindications to MR scanning including, pregnancy, weight inappropriate for height, ferrous objects within the body (only for the sub-sample asked to undergo fMRI.)

Exclusion Criteria:

Exclusion Criteria

* Acute or progressive cardiac, vascular, renal, respiratory, neurological disorders or malignancy.
* Active psychiatric diagnosis or psychological condition, or active drug/alcohol abuse.
* Lower motor neuron damage or radiculopathy.
* Orthopedic impairment. **
* More than one stroke.
* Cerebellar dysfunction.
* Fugl-Meyer lower limb motor sub-score greater than 32.
* No simultaneous gait rehabilitation participation.
* Pregnant.
* Claustrophobia (only for the sub-sample asked to undergo fMRI.)
* Criteria specific to MR scanning, including pregnancy, weight inappropriate for height, ferrous objects within the body (only for the sub-sample asked to undergo fMRI.)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janis J. Daly, PhD MS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened out if presenting with unstable medical conditions that could affect safety.
Groups:
- Gait and Cognitive Training: Gait rehabilitation combined with cognitive rehabilitation
- Gait and Arm Training: Gait rehabilitation combined with arm (reach/grasp) rehabilitation
Period: Overall Study
Arm/Group | Gait and Cognitive Training | Gait and Arm Training
Started | 5 | 7
Completed | 4 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gait and Cognitive Training | Gait and Arm Training | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in the Gait Assessment and Intervention (G.A.I.T.) Score
Description: Coordination of walking, scored using the investigators' novel G.A.I.T. measure. This measure evaluated limb and joint movements while participants walk overground at preferred speed. Range of scale: 0 (normal) to 64 (extremely discoordinated gait).
Time Frame: pre-training (0 weeks), post training (about 12 weeks)
Population: Adults with chronic post-stroke hemiparesis and gait deficits
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gait and Cognitive Training | Gait and Arm Training
Number analyzed (Participants) | 4 | 7
units on a scale
  pre treatment mean | 28.8 (6.9) | 29.5 (3.8)
  post treatment mean | 29.9 (5.9) | 28.7 (7.7)
Statistical Analysis 1: Comparison: Gait and Cognitive Training vs Gait and Arm Training; Test type: Superiority; p = 0.54, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Gait and Cognitive Training | Gait and Arm Training
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 1/4 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gait and Cognitive Training (N=4) | Gait and Arm Training (N=7)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early closure leading to small numbers of subjects analyzed. early enrollment closure due to inability for the institution to hire skilled clinicians in a timely manner in order to enroll and treat participants in the available time frame.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes